CLINICAL TRIAL: NCT01861886
Title: A Multi-Centre Clinical Study to Evaluate the Safety and Effectiveness of the ESS505® Device to Prevent Pregnancy in Women Who Are Seeking Permanent Contraception
Brief Title: The Safety and Effectiveness of the Essure (Model ESS505) Device to Prevent Pregnancy in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16972; ESS505-003 (Other: Company Internal)
Record Dates: First submitted 2013-02-20; First posted 2013-05-24 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Contraception
Keywords: Birth control; Permanent Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ESS505 (Experimental): Bilateral hysteroscopic placement of the permanent birth control system, Model ESS505 in the proximal portion of the fallopian tubes using a transvaginal approach. Subsequent transvaginal ultrasound (TVU) or hysterosalpingogram (HSG) was performed approximately ≤ 3 hours and 90 days following insert placement.
  Interventions: Device: ESS505 (BAY1454033)

INTERVENTIONS:
Device: ESS505 (BAY1454033) — Bilateral hysteroscopic placement of the permanent birth control system, Model ESS505 in the proximal portion of the fallopian tubes using a transvaginal approach. Subsequent transvaginal ultrasound (TVU) or hysterosalpingogram (HSG) was performed approximately ≤ 3 hours and 90 days following insert placement.

SUMMARY:
To evaluate the safety and long-term (approximately one year) effectiveness of the Essure System for Permanent Birth Control ESS505 device in preventing pregnancy.

DETAILED DESCRIPTION:
This study has previously been posted by Conceptus, Inc. After acquiring Conceptus, Inc., Bayer is now the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Female with age range 21 to 44 years
* Subjects who are seeking permanent contraception
* Subjects with body weight within range of 40 - 136 kilograms (90-300 pounds)
* Subjects willing to accept the risk of pregnancy occurring while relying solely on the ESS505 as contraception
* Subjects for whom medical history and physical examination indicates bilateral viable and patent fallopian tubes
* Subjects who are able to comply with the protocol required follow-up visits (e.g., 3 month clinic visit, and the 12-month telephone interview)
* Subjects who provide written informed consent prior to enrolment
* Subjects who have sufficient mental capability to provide clinically relevant and reliable feedback regarding her experience wearing the device
* Subjects agrees that her anonymised personal data will be made available to Study sponsor, requisite regional and international regulatory bodies
* Subjects for whom there are no contraindications for use as described in the ESS505 Instructions for Use (IFU)

Exclusion Criteria:

* Subjects with known proximal tubal occlusion in either fallopian tube
* Subjects who have undergone fallopian tube sterilization procedure
* Subjects diagnosed with unicornuate uterus
* Subjects diagnosed with endometrial or myometrial pathology which may prevent fallopian tube ostia assessment
* Subjects scheduled to undergo concomitant intrauterine procedures at the time of ESS505 placement; IUD removal is not considered a concomitant procedure
* Subjects suspected of being or confirmed pregnant
* Subjects post-partum or has undergone pregnancy termination ≤6 weeks of scheduled ESS505 placement
* Subjects diagnosed with active upper or lower pelvic infection
* Subjects for whom there are one or more contraindications for use as described in the ESS505 IFU
* Subjects have positive pre-procedure pregnancy test

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2013-12-19 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of confirmed pregnancy at 3 months among successful bilateral implant subjects relying solely on the ESS505 for contraception. | 3 months

SECONDARY OUTCOMES:
Occurrence of confirmed pregnancy at 12 months among successful bilaterally implant subjects relying solely on the ESS505 for contraception | 12 months
Frequency (number) of reported ESS505 placement procedure-related AEs | 3 months
  Date of enrollment, 31 JAN 2013 to data cut-off for this interim CSR, 23 FEB 2014.
Severity of reported ESS505 placement procedure-related AEs | 3 months
  31 JAN 2013 to data cut-off for this interim CSR, 23 FEB 2014
Frequency (number) of reported ESS505 (device) wearing-related AEs | 3 months
  31 JAN 2013 to data cut-off for this interim CSR, 23 FEB 2014
Severity of reported ESS505 wearing-related AEs | 3 months
  31 JAN 2013 to data cut-off for this interim CSR, 23 FEB 2014

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Netherlands (4):
  - Hoofddorp
  - Nieuwegein
  - Tiel
  - Zwolle
- Córdoba, Córdoba, Spain